CLINICAL TRIAL: NCT05823623
Title: A Phase II Single-arm Clinical Trial of Inetetamab Combined With Pyrotinib Plus Oral Vinorelbine for the Treatment of Patients With HER2-positive Metastatic Breast Cancer
Brief Title: Inetetamab Combined With Pyrotinib Plus Oral Vinorelbine for the Treatment of HER2-positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-494
Record Dates: First submitted 2023-03-23; First posted 2023-04-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab combined with Pyrotinib plus Oral Vinorelbine (Experimental): Inetetamab: 8mg/kg for the first dose, 6mg/kg for the following doses, intravenous, every 3 weeks for one cycle. Pyrotinib: 400mg, oral, every day. Vinorelbine: 60mg/m2, oral, every week.
  Interventions: Drug: Inetetamab; Drug: Pyrotinib; Drug: Oral Vinorelbine Tartrate

INTERVENTIONS:
Drug: Inetetamab — Patients with HER2-positive metastatic breast cancer after progression on trastuzumab are enrolled and receive treatment.
Drug: Pyrotinib — Patients with HER2-positive metastatic breast cancer after progression on trastuzumab are enrolled and receive treatment.
Drug: Oral Vinorelbine Tartrate — Patients with HER2-positive metastatic breast cancer after progression on trastuzumab are enrolled and receive treatment.

SUMMARY:
In this phase 2 single-arm clinical trial, 30 patients with HER2-positive metastatic breast cancer after progression on trastuzumab are enrolled and receive treatment of Inetetamab plus Pyrotinib plus Oral Vinorelbine. The study aimed to access the efficacy and safety of Inetetamab combined with Pyrotinib and Oral Vinorelbine in HER2-positive metastatic breast cancer patients after progression on trastuzumab.

DETAILED DESCRIPTION:
Trastuzumab is an important agent for the treatment of patients with HER2-positive metastatic breast cancer. However, a considerable number of patients will develop resistance to trastuzumab treatment. Previous studies have shown that multiple mechanisms mediate trastuzumab resistance, such as abnormal extracellular domain of the HER2 receptor, HER3 mutation and activation of bypass signaling pathway. To overcome these resistance mechanisms, the combination of trastuzumab with HER2-targeting tyrosine kinase inhibitor (TKI) is an effective strategy. In this phase 2 single-arm clinical trial, 30 patients with HER2-positive metastatic breast cancer after progression on trastuzumab are enrolled and receive treatment of Inetetamab plus Pyrotinib plus Oral Vinorelbine. The study aimed to access the efficacy and safety of Inetetamab combined with Pyrotinib and Oral Vinorelbine in HER2-positive metastatic breast cancer patients after progression on trastuzumab. The primary end point is Progressive-free Survival (PFS). The secondary end points are Overall Survival (OS), Overall Response Rate (ORR), Clinical Benefit Rate (CBR) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Aged ≥ 18 years.
2. Metastatic breast cancer confirmed by pathology or imaging.
3. Pathological diagnosis of HER2 positive (definition: immunohistochemical (IHC) 3+, or IHC 2+ with in situ hybridization (ISH) testing of amplification.
4. Previously received trastuzumab treatment.
5. At least one Measurable target lesion according to RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) score 0- 2.
7. Sufficient organ function: Neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L, Platelet count (PLT) ≥ 100 × 10 ^ 9 / L, hemoglobin (Hb) ≥90 g/L，total bilirubin (TBIL) ≤ 1.5 × upper limit of normal value (ULN), alanine aminotransferase (ALT / AST) ≤ 2.5 × ULN (liver metastasis patients ≤ 5×ULN), serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60 ml/min, Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

1. Allergic to the ingredients of the study drug.
2. Symptomatic brain or meningeal metastasis.
3. Gastrointestinal dysfunction or gastrointestinal diseases (including active ulcers).
4. LVEF <50%; clinical manifestations of patients with obvious arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency, and severe valvular disease.
5. Any other medical, social or psychological conditions which are inappropriate to participate in this trial.
6. Pregnant or lactating women, women of childbearing age who refused to take effective contraceptive measures during the study period.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival，PFS | 2 years
  The time from the beginning of treatment to the progression or death of the patient

SECONDARY OUTCOMES:
overall survival，OS | 4 years
  The time from the beginning of treatment to the death of the patient
Objective Response Rate，ORR | 2 year
  The percentage of participants whose best overall response, according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, is either complete response (CR) or partial response (PR)
Clinical Benefit Rate，CBR | 2 year
  the percentage of participants whose best overall response, is either CR, PR or stable disease (SD) lasting for at least 24 weeks
adverse events | 2 years
  The probability and severity of adverse reactions related to the treatment were assessed by CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v5.0.

OTHER OUTCOMES:
Exploration of biomarkers | 1 year
  To explore the potential biomarkers for the efficacy of combined therapy. The biomarkers will be tested by next-generation sequence

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Huang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin N, Xu Y, Wang S, Sun C, Yan X, Yang F, Liang Y, Chen W, Huang X. Inetetamab combined with pyrotinib and oral vinorelbine for patients with human epidermal growth factor receptor 2 positive advanced breast cancer: A single-arm phase 2 clinical trial. Cancer Pathog Ther. 2023 Oct 30;2(1):31-37. doi: 10.1016/j.cpt.2023.10.004. eCollection 2024 Jan. PMID 38328709